CLINICAL TRIAL: NCT04585997
Title: How to "Choosebetweenamab" for Severe Asthma, Comparing Treatment With Mepolizumab and Omalizumab for Patients With Severe Allergic and Eosinophilic Asthma.
Brief Title: Comparing Treatment Efficacy With Mepolizumab and Omalizumab in Severe Asthma - "Choosebetweenamab".
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Newcastle, Australia (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Professor Peter Wark, Professor and Senior Staff Respiratory Specialist, University of Newcastle, Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/08/15/3.01
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Asthma; Eosinophilic Asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab; Omalizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: People assessing outcomes and analyzing results are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepolizumab (Active Comparator): Mepolizumab
  Interventions: Drug: Mepolizumab
- Omalizumab (Active Comparator): Omalizumab
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab 100mg subcutaneous injection monthly for 6 months
  Other Names: Nucala
  Arms: Mepolizumab
Drug: Omalizumab — Omalizumab subcutaneous injection every 2-4 weeks (dosage determined by the Omalizumab nomogram).
  Other Names: Xolair
  Arms: Omalizumab

SUMMARY:
Mepolizumab is an anti-interleukin-5 ( IL-5) monoclonal antibody that neutralizes IL-5 and reduces eosinophil counts in both sputum and blood. Omalizumab is an anti-immunoglobulin E (IgE) monoclonal antibody (mAb) used in the treatment of severe allergic eosinophilic asthma

The investigators propose that in patients with the dual phenotypes of severe allergic and eosinophilic asthma, that Mepolizumab is as effective as Omalizumab. However, this trial will also identify key clinical biomarkers that will clarify which patients will respond best to each of these interventions.

This study will be the first direct clinical comparison of these agents and will apply expert clinical characterization, along with cutting edge biotechnology to better inform treatment choices for severe asthma. This is an important and urgent management problem facing the Australian pharmaceutical scheme, where imprecision in prescribing will result in reduced clinical effectiveness as well as substantial and sustained costs.

DETAILED DESCRIPTION:
'Choosebetweenamab' will compare active treatment arms (Mepolizumab and Omalizumab) for efficacy and adverse events in a Phase 4, parallel arm, randomized controlled trail setting with computer generated randomization (permuted block randomization, with block sizes of 4 or 6, stratified by baseline eosinophil count using a median split). There is no placebo control. Particpants will not be blinded but masking will be used for people assessing outcomes and analyzing data.

'Chossebetweenamab' will also include a secondary outcome substudy (ISS 11066) to assess biomarkers of efficacy response to treatment using single cell sequencing of peripheral blood cells. Blood samples are taken from the randomized patients in each treatment arm (Mepolizumab and Omalizumab) at baseline and gene expression changes assessed using transcriptomic single cell sequencing of patient white blood cells. The data generated from this will be compared to the clinical outcomes of 'Choosebetweenamab' at all follow-up time points. Single cell gene expression and cell type cluster patterning will be compared to the primary and secondary outcomes to identify baseline predictors (gene and cell type) of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a duration of asthma of greater than one year.
* They must have confirmed asthma defined as: (i) forced expiratory volume (FEV1) reversibility greater than or equal to 12%, and greater than or equal to 200 mL at baseline within 30 minutes after administration of salbutamol (200 to 400 micrograms), or (ii) airway hyperresponsiveness defined as a greater than 20% decline in FEV1 during a direct bronchial provocation test or greater than 15% decline during an indirect bronchial provocation test, or (iii) peak expiratory flow (PEF) variability of greater than 15% between the two highest and two lowest peak expiratory flow rates during 14 days.
* They must have evidence of poor asthma control despite optimal ICS and long acting beta agonist (LABA), be treated by a respiratory physician or immunologist, and have demonstrated acceptable adherence and inhaler technique. Poor control is defined as: evidence of an FEV1 <80% of predicted in the last year on at least one occasion; treatment with OCS, either daily for at least 6 weeks, or a cumulative dose of OCS of at least 500 mg prednisolone equivalent in the previous 12 months, unless contraindicated or not tolerated.
* In addition they must demonstrate an: (a) an Asthma Control Questionnaire (ACQ-5)38 score of at least 2.0, as assessed in the previous month, and (b) while receiving optimised asthma therapy in the past 12 months, experienced at least 1 admission to hospital for a severe asthma exacerbation, or 1 severe asthma exacerbation, requiring documented use of OCS initiated or increased for at least 3 days, or parenteral corticosteroids prescribed/supervised by a physician.
* They must also demonstrate evidence of a dual allergic/ eosinophilic phenotype. This is defined as: a total serum IgE >30IU/mL, past or current evidence of atopy documented by skin prick testing or radioallergosorbent assay, and the participant must have a blood eosinophil count greater than or equal to 300 cells per microlitre in the last 6 weeks.

Exclusion Criteria:

* Do not fulfil inclusion criteria
* Unable to attend appointments
* Significant psychiatric illness

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-11-03 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
ACQ5 | Assessed after 6 months treatment
  The primary outcome will be Asthma control questionairre (ACQ)5, adjusted for baseline ACQ5

SECONDARY OUTCOMES:
Exacerbations | every month up to 6 months after treatment commenced
  Number of Exacerbations, requiring change in oral corticosteroids, with either a course of prednisone for at least 3 days, or in those on regular OCS an increase in dose of at least 50% for at least 3 days. Patient reported monthly
Time to first exacerbation reported, by patient or health provider | every month up to 6 months after treatment commenced
  Time to first exacerbation reported, by patient or health provider
Hospital admissions | every month up to 6 months after treatment commenced
  Number of admissions to hospital patient reported
Oral corticosteroids | every month up to 6 months after treatment commenced
  Reduction in dose of regular OCS, confirmed by health care provider and patient reported
Spirometry | every month up to 6 months after treatment commenced
  Change in spirometry, FEV1., measured at time treatment commences and 6 months after treatment
Continuing treatment | 6 months post intervention
  Proportion continuing on Australian PBS treatment (successful treatment). The number at the conclusion of the 6 months that will continue treatment. reported by health provider
Adverse events | every month up to 6 months after treatment commenced
  Adverse events; i.e. injection site reaction, reported. Headaches, reported, rash, reported, allergic reaction, reported. Any other relevant adverse event report. Patient and health care provider reported
Emergency department presentation | every month up to 6 months after treatment commenced
  Number of emergency department presentations, patient and health care provider reported
Overall dose of oral corticosteroids | 6 months post intervention
  Overall dose of systemic corticosteroids used during the 6 months after treatment commences. Patients and health care provided
Change in gene expression measured by single cell RNA sequencing of peripheral blood cells (ISS 11066) | Measured prior to treatment and clinical outcomes at 6 months after treatment
  ISS 11066 is a substudy of Choosebetweenamab using transcriptomic single cell sequencing of patient white blood cells from both treatment groups at baseline. The data generated from this will be compared to the above clinical outcomes at all follow-up time points. Single cell gene expression and cell type cluster patterning delineated through bioinformatic data processing will be inputted with clinical outcomes into a GLM to identify baseline predictors (gene and cell type) of treatment effect

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wark, MBBS/PhD, Principal Investigator — University of Newcastle and Hunter New England Health
Locations (1):
- John Hunter Hospital, New Lambton, New South Wales, Australia

DOCUMENTS (2):
  • Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT04585997/ICF_000.pdf
  • Study Protocol (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT04585997/Prot_001.pdf